CLINICAL TRIAL: NCT04174118
Title: A Phase 1 Single Ascending Dose, Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics Study of Subcutaneously Administered Belcesiran in Healthy Adult Volunteers
Brief Title: Study of DCR-A1AT in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dicerna Pharmaceuticals, Inc., a Novo Nordisk company (Industry)
Responsible Party: Sponsor
Organization: Novo Nordisk A/S (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: DCR-A1AT-101
Record Dates: First submitted 2019-11-06; First posted 2019-11-22 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-09

CONDITIONS: Alpha 1-Antitrypsin Deficiency
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- belcesiran (Experimental): Healthy volunteers will be administered a single dose of belcesiran.
  Interventions: Drug: belcesiran
- Placebo (Placebo Comparator): Healthy volunteers will be administered a single dose of matching placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: belcesiran — belcesiran will be administered subcutaneously (SC) at dose levels planned.
  Arms: belcesiran
Drug: Placebo — Sterile normal saline (0.9% NaCL) matching volume of belcesiran doses will be administered subcutaneously (SC).
  Arms: Placebo

SUMMARY:
This is a research study to test an experimental study drug (belcesiran, also known as DCR-A1AT). This drug is being tested to see if it helps people with a rare condition known as Alpha-1 Antitrypsin Deficiency, or A1ATD. Prior to initiation of this study belcesiran had not yet been tested in humans. All study participants will be randomly assigned to either receive the study drug or a placebo. This will allow for the sponsor to compare the effects of the study drug with that of the placebo. A placebo looks like the study drug but does not contain any of the study drug.

The main purpose of the first part of the study is to evaluate the safety profile of the study drug in people who do not have A1ATD. This part of the study will also help find the dose of the study drug that has an acceptable safety profile for testing.

DETAILED DESCRIPTION:
A1ATD- associated liver disease is a progressive Alpha-1 Antitrypsin-Deficiency Associated Liver Disease condition resulting in liver fibrosis, cirrhosis, and hepatocellular carcinoma. The lack of functional A1AT in individuals with PiZZ genotype, in conjunction with other precipitating factors, can lead to unchecked activity in neutrophil elastases in the alveoli; causing emphysema and chronic obstructive pulmonary disease (COPD). This loss-of-function mechanism can be addressed with intravenous augmentation therapy, which aims to substitute the missing A1AT by infusing alpha1 proteinase inhibitor (A1PI), purified from pooled human plasma.

While augmentation therapy can address the loss of A1AT in the lungs, no treatment exists for the associated liver disease.

Given the severity of the disease, with approximately 10% of affected patients developing liver cirrhosis and a subgroup of those patients in need of liver transplantation, and lack of an effective treatment that addresses the toxic hepatic "gain-of-function" mechanism, there is an urgent unmet medical need to develop a therapy that can help in this particular patient population.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female aged 18 to 55 years, inclusive. Female participants must be either surgically sterile or postmenopausal. No women of childbearing potential are eligible for enrollment.
* Overtly Healthy, as determined by the investigator.
* Serum A1AT protein concentration >100 mg/dL
* Adequate forced expiratory volume in one second (FEV1) and adequate FEV1/forced vital capacity (FVC) ratio
* Non-smokers with a <2 pack-year history and smoking cessation for at least 6 months with a negative urinary cotinine test a screening

Exclusion Criteria:

* Presence of any condition or comorbidities that would interfere with study compliance or data interpretation or potentially affect participant safety
* Clinically significant abnormal laboratory tests
* Received an experimental drug within past 4 months
* Prior to use of RNAi drug or oligonucleotide-based therapy
* Known human immunodeficiency virus (HIV), hepatitis C virus (HCV), or Hepatitis B (HBV)
* Serum creatinine or estimated glomerular filtration rate (eGFR) outside normal reference ranges.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-10-24 (Actual); Primary Completion 2021-07-06 (Actual); Study Completion 2023-03-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | approximately up to 2 months
  The incidence of adverse events (AE), serious adverse events (SAE), DLT, and AE leading to study drug discontinuation
Evaluating safety and tolerability through physical exams | approximately up to 2 months
  The incidence of clinically significant physical examination (PE) findings
Changes in 12-lead electrocardiograms (ECG) | approximately up to 2 months
  Absolute QTc > 500 msec and/or QTc change of > 60 msec from baseline will be evaluated

SECONDARY OUTCOMES:
Urine pharmacokinetics (PK) of belcesiran | up to Day 3
  Maximum observed concentration (Cmax)
Plasma pharmacokinetics (PK) of belcesiran | up to 57 days
  Maximum observed concentration (Cmax)
Plasma pharmacokinetics (PK) of belcesiran | up to 57 days
  Area under the curve (AUC)
Urine pharmacokinetics (PK) of belcesiran | up to Day 3
  Area under the curve (AUC)
Urine pharmacokinetics (PK) of belcesiran | up to Day 3
  Minimum observed concentration (Cmin)
Plasma pharmacokinetics (PK) of belcesiran | up to 57 days
  Minimum observed concentration (Cmin)
Plasma pharmacokinetics (PK) of belcesiran | up to 57 days
  Time to maximum concentration (Tmax)
Urine pharmacokinetics (PK) of belcesiran | up to Day 3
  Time to maximum concentration (Tmax)
Urine pharmacokinetics (PK) of belcesiran | up to Day 3
  Terminal elimination half-life (t1/2)
Plama pharmacokinetics (PK) of belcesiran | up to 57 days
  Terminal elimination half-life (t1/2)
Change in protein concentration | up to day 57
  Changes in A1AT protein concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bowman, MD, Study Director — Dicerna Pharmaceuticals
Locations (2):
- Auckland Clinical Studies, Grafton, Auckland, New Zealand
- Clinical Trial Consultants AB, Uppsala, Sweden

REFERENCES:
- [Derived] Remih K, Amzou S, Strnad P. Alpha1-antitrypsin deficiency: New therapies on the horizon. Curr Opin Pharmacol. 2021 Aug;59:149-156. doi: 10.1016/j.coph.2021.06.001. Epub 2021 Jul 10. PMID 34256305